CLINICAL TRIAL: NCT05813405
Title: Study on Integration of Cardiovascular and Cerebrovascular Diseases
Brief Title: Correlation Between Coronary Artery and Brain Study
Status: Not yet recruiting | Type: Observational
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Xin Lou, Deputy Director of Department of Radiology, Chinese PLA General Hospital
Other Study IDs: Heart-Brain Correlation-301
Record Dates: First submitted 2023-04-03; First posted 2023-04-14 (Actual); Last update posted 2023-04-14 (Actual); Status verified 2023-04

CONDITIONS: Cardiovascular and Cerebrovascular Diseases
Keywords: Cardiovascular disease; Cerebrovascular disease; Intervention treatment; multimodal imaging technology
MeSH Terms: conditions — Cerebrovascular Disorders; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Experimental: Antihypertensive therapy Hypotension and improved ventilation treatment Intervention treatment for other risk factors — Experimental: Antihypertensive therapy Hypotension and improved ventilation treatment Intervention treatment for other risk factors

SUMMARY:
To explore the pathogenesis of cardiovascular and cerebrovascular diseases through study on cardio-cerebral integration based on multimodal imaging technology, and clinical evaluation of its secondary diseases and intervention treatment.

Cardiovascular and cerebrovascular diseases are leading causes of death and disability worldwide. Atherosclerosis of the large arteries of the brain and the heart has received extensive attention and in-depth research. By contrast, the epidemiology of small-vessel disease (SVD) of the brain and heart is less well established.

The vascular anatomy of the heart and brain is similar in that conduit arteries are distributed on the surface of these organs with tissue perfusion achieved through deep penetrating arteries. In the heart, SVD involves the deep penetrating coronary arterioles and the subendocardial plexus of microvessels. The clinical sequelae of SVD in the heart include stable and acute coronary syndromes and heart failure in the longer term. SVD in the brain mainly involves small subcortical arterioles. If a vascular occlusion occurs, small lacunar lesions can occur, while long-term chronic ischemia caused by SVD may manifest as vascular cognitive impairment. There is a close relationship between cardiovascular and cerebrovascular diseases, and cardiovascular risk factors are related to the etiology of cerebral SVD. However, whether this relationship has a causal remains unclear.

Thus, the study of cardiovascular and cerebrovascular integration based on multimodal imaging technology has important value for the diagnosis, efficacy evaluation, and prognosis judgment of cardiovascular and cerebrovascular diseases.

DETAILED DESCRIPTION:
Patients:

Patients with heart disease, such as coronary heart disease, atrial fibrillation or flutter, cardiac insufficiency, etc. were included. And collect the patient's brain MRI data simultaneously. To explore the relationship between embolic properties and cerebral embolism, the relationship between cardiovascular and cerebrovascular diseases and cognitive dysfunction, and also comparison of changes in cardiocerebral structure and function before and after intervention with risk factors.

Imaging protocols:

Brain magnetic resonance acquisition: Use a 3.0T magnetic resonance scanner for imaging, and the acquisition coil uses a dedicated brain coil. The scan sequence includes routine T1WI, T2WI, FLAIR, and other sequences. If necessary, further patient functional magnetic resonance examinations such as BOLD, 3D T2FLAIR, 3D FSPGR-T1WI, 3D pCASL, DTI, and 3D SWI are performed.

Cardiac magnetic resonance acquisition: cardiac and coronary CTA, cardiac and coronary MRA; Myocardial perfusion magnetic resonance imaging, etc.

Treatment:

Intervention treatment for risk factors

Follow-up:

Baseline (MRI+clinical evaluation); 3-months, 6-months,1-year (MRI+clinical evaluation).

ELIGIBILITY:
Inclusion Criteria:

① Patients with cardiovascular diseases such as coronary heart disease, cardiac dysfunction, arrhythmia, precordial pain, and patients with atrial fibrillation or atrial flutter have not received anticoagulant treatment Meet the diagnostic criteria for hypertension; ③ Meet the diagnostic criteria for obstructive sleep apnea hypopnea syndrome; ④ No history of craniocerebral injury; ⑤ No neuropsychiatric diseases.

Exclusion Criteria:

① Routine MRI examination found that there were significant lesions in the heart and brain that affected the structure of the heart and brain Patients who cannot tolerate MRI examination.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cardiovascular and cerebrovascular diseases patients
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-04-03 (Estimated); Primary Completion 2028-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
To Study the relationship between the nature of left atrial thrombus and cardiogenic cerebral infarction | 5 year
To evaluate changes in brain structure and function in patients with cardiovascular and cerebrovascular diseases, and analyze the relationship between cardiovascular and cerebrovascular diseases and cognitive impairment | 5 year
To evaluate the impact of risk factor intervention on the structure and function of heart and brain in patients with cardiovascular and cerebrovascular diseases | 5 year
  Myocardial MRI perfusion and 3D pCASL sequence will be used to assess the cardiac and cerebral perfusion in each treated patient before and after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Xin Lou, MD/PhD, Study Chair — Chinese PLA General Hospital